CLINICAL TRIAL: NCT05280314
Title: Phase II, Multi-cohort Trial of Neoadjuvant and Post-surgery IO102-IO103 and Pembrolizumab KEYTRUDA® in Patients With Selected Resectable Tumors
Brief Title: Phase II Trial of Neoadjuvant and Adjuvant IO102-IO103 and Pembrolizumab KEYTRUDA® in Patients With Resectable Tumors
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: IO Biotech (Industry)
Collaborators: Theradex (Industry); Almac (Industry); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IO102-IO103-032/IOB-032; MK-3475-E40 (Other: Merck Sharp & Dohme LLC.)
Record Dates: First submitted 2022-02-22; First posted 2022-03-15 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Melanoma; Squamous Cell Carcinoma of Head and Neck
MeSH Terms: conditions — Melanoma; Squamous Cell Carcinoma of Head and Neck | interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: Multicenter, Multi-arm, Two indications, One Cohort SCCHN 2 Cohorts melanoma (1 cohort randomized and one cohort not randomized)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort A - Melanoma (Experimental): Cutaneous resectable Stage III melanoma.
  Neoadjuvant Treatment (3 cycles): Subcutaneous IO102-IO103 (IO102 85 μg and IO103 85 μg) and intravenous Pembrolizumab KEYTRUDA® 200mg Q3W.
  Post-surgery Treatment (15 cycles): Subcutaneous IO102-IO103 (IO102 85 μg and IO103 85 μg) and intravenous Pembrolizumab KEYTRUDA® 200mg Q3W.
  Interventions: Drug: IO102-IO103; Drug: Pembrolizumab KEYTRUDA®
- Cohort B - SCCHN (Experimental): Stage III or IVA resectable locoregionally advanced Squamous cell carcinoma of the head and neck (SCCHN) of the oral cavity, oropharynx (HPV-negative), hypopharynx, or larynx
  Neoadjuvant Treatment (2-3 cycles): Subcutaneous IO102-IO103 (IO102 85 μg and IO103 85 μg) and intravenous Pembrolizumab KEYTRUDA® 200mg Q3W Post-surgery Treatment (15 cycles): Subcutaneous IO102-IO103 (IO102 85 μg and IO103 85 μg) and intravenous Pembrolizumab KEYTRUDA® 200mg Q3W.
  Interventions: Drug: IO102-IO103; Drug: Pembrolizumab KEYTRUDA®
- Cohort C (Experimental): Cutaneous resectable Stage III melanoma. Neoadjuvant Treatment (3 cycles): Subcutaneous IO102-IO103 (IO102 85 μg and IO103 85 μg) and intravenous Pembrolizumab KEYTRUDA® 200mg Q3W (Arm A) versus intravenous Pembrolizumab KEYTRUDA® 200mg Q3W alone (Arm B) Post-surgery Treatment (15 cycles): Subcutaneous IO102-IO103 (IO102 85 μg and IO103 85 μg) and intravenous Pembrolizumab KEYTRUDA® 200mg Q3W (Arm A) versus Pembrolizumab KEYTRUDA® 200mg Q3W alone (Arm B)
  Interventions: Drug: IO102-IO103; Drug: Pembrolizumab KEYTRUDA®

INTERVENTIONS:
Drug: IO102-IO103 — IO102-IO103 is a combination of an indoleamine 2,3-dioxygenase 1 (IDO1) peptide (IO102) and a programmed death-ligand 1 (PD-L1) peptide (IO103), emulsified with an adjuvant (Montanide ISA 51 VG).
Drug: Pembrolizumab KEYTRUDA® — Pembrolizumab KEYTRUDA® administered intravenously

SUMMARY:
This is a multicenter, multi-arm trial evaluating anti-tumor activity, safety, and immune infiltration of IO102-IO103 in combination with pembrolizumab KEYTRUDA® as neoadjuvant and post-surgery treatment. This proof-of-concept trial will include patients with resectable tumors in at least 2 indications.

DETAILED DESCRIPTION:
This is a multicenter, multi-arm trial evaluating anti-tumor activity, safety, and immune infiltration of IO102-IO103 in combination with pembrolizumab KEYTRUDA® as neoadjuvant and post-surgery treatment. Approximately 60 patients with melanoma or SCCHN will be included (approximately 15 for each indication).During the neoadjuvant period, patients in cohort A, cohort B and Cohort C (Arm A) will receive IO102-IO103 and pembrolizumab KEYTRUDA® Q3W. Patients in Cohort C (Arm B) will receive pembrolizumab KEYTRUDA® Patients with melanoma will receive 3 doses of neoadjuvant treatment. Patients with SCCHN will receive 2 or 3 doses of neoadjuvant treatment, at the investigator's discretion. Surgical resection will be performed 1 to 3 weeks after the last dose of neoadjuvant treatment. All patients in cohort A,B and Cohort C (Arm A)will receive post-surgery treatment with IO102-IO103 and pembrolizumab KEYTRUDA® for a total of 15 cycles (up to 45 weeks). Patients in Cohort C (Arm B) will receive post-surgery treatment with pembrolizumab KEYTRUDA® for a total of 15 cycles (up to 45 weeks).

Patients with melanoma and patients with SCCHN who do not require SOC RT ± cisplatin will start post-surgery treatment after adequate recovery from surgery (approximately 1 to 2 months; no more than 12 weeks).Patients with SCCHN who require postoperative SOC therapy after surgery will start post-surgery IO102-IO103 and pembrolizumab KEYTRUDA® after adequate recovery from SOC therapy (approximately 1 to 2 months; no more than 12 weeks).

Objective response will be based on imaging; pathologic tumor response of the surgical specimens will be assessed at the time of surgery. Safety will be assessed by recording adverse events. The primary endpoint will be the percentage of patients with major pathologic response (MPR) in the resected tumor tissue after neoadjuvant treatment. Secondary endpoints include disease-free survival (DFS) at 2 years after surgery. All patients will have an end-of-treatment visit approximately 4 weeks after their last dose of trial treatment. Follow-up visits will be conducted at 6 and 12 months after the end-of-treatment visit. Following completion of the 12-month follow-up period, long-term follow-up for overall survival (OS) will be conducted every 6 months for at least a further 12 month.

ELIGIBILITY:
Melanoma-specific inclusion criteria:

• Histologically or cytologically confirmed diagnosis of cutaneous stage III melanoma according to the American Joint Committee on Cancer (AJCC) 8th edition.

Patients with resectable tumors are eligible for this trial either at presentation for primary melanoma with concurrent regional nodal metastasis or at the time of clinically detected nodal recurrence; they may belong to any of the following groups:

* Primary cutaneous melanoma with clinically apparent regional lymph node metastases
* Clinically detected recurrent melanoma at the proximal regional lymph node(s) basin
* Clinically detected primary cutaneous melanoma involving multiple regional nodal groups
* Clinically detected nodal melanoma (if single site) arising from an unknown primary
* Relapsed resectable stage III melanoma

SCCHN-specific inclusion criteria:

• Stage III or IVA resectable locoregionally advanced SCCHN of the oral cavity, oropharynx (with known HPV-negative or p16-negative status assessed per institution standard or centrally), hypopharynx, or larynx.

Inclusion criteria applicable across cohorts:

In addition to the indication-specific inclusion criteria, a patient must meet all the following general criteria to be eligible for participation in this trial:

1. Measurable disease based on Response Evaluation Criteria In Solid Tumors (RECIST) 1.1
2. Candidate for surgical resection with curative intent
3. The patient (or legally acceptable representative if applicable) provides written informed consent for the trial.
4. Age ≥18 years on the day of signing the informed consent form
5. Have provided archival tumor tissue sample or newly obtained core or excisional biopsy of a tumor lesion not previously irradiated. Formalin-fixed, paraffin embedded (FFPE) tissue blocks are preferred to slides.
6. Eastern Cooperative Oncology Group (ECOG) performance score status of 0 or 1
7. Adequate organ function as defined below performed on screening labs obtained within 4 weeks before first dose:

   * Absolute neutrophil count (ANC) ≥1500/µL
   * Platelets ≥100 000/µL
   * Hemoglobin ≥9.0 g/dL or ≥5.6 mmol/L (Note: Criterion must be met without packed red blood cell transfusion within the prior 2 weeks. Patients can be on stable dose of erythropoietin [≥ approximately 3 months].)
   * Creatinine or measured or calculated creatinine clearance (glomerular filtration rate can also be used in place of creatinine or creatinine clearance) ≤1.5 × upper limit of normal (ULN) or ≥30 mL/min for patient with creatinine levels >1.5 × institutional ULN
   * Serum total bilirubin ≤1.5 × ULN or direct bilirubin ≤ ULN for patients with total bilirubin levels >1.5 × ULN
   * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 × ULN
   * International normalized ratio (INR) or prothrombin time (PT) ≤1.5 × ULN unless the patient is receiving anticoagulant therapy as long as PT or partial thromboplastin time (PTT) is within the therapeutic range of intended use of anticoagulants
   * Activated partial thromboplastin time (aPTT) ≤1.5 × ULN unless the patient is receiving anticoagulant therapy as long as PT or PTT is within the therapeutic range of intended use of anticoagulants
8. Women of childbearing potential: Negative urine or serum pregnancy within 72 hours prior to receiving the first dose of trial medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
9. Women of childbearing potential: Willing to use highly effective contraception or abstain from heterosexual activity for the duration of the trial and for at least 120 days after the last dose of trial medication
10. HIV-infected patients must be on anti-retroviral therapy (ART) and have a well-controlled HIV infection/disease defined as:

a Patients on ART must have a CD4+ T-cell count >350 cells/mm3 at time of screening b Patients on ART must have achieved and maintained virologic suppression defined as confirmed HIV RNA level below 50 copies/mL or the lower limit of qualification (below the limit of detection) using the locally available assay at the time of screening and for at least 12 weeks prior to first dose of trial medication (Day 1) c Patients on ART must have been on a stable regimen, without changes in drugs or dose modification, for at least 4 weeks prior to first dose of trial medication (Day 1) 11. Patients who are hepatitis B surface antigen (HBsAg) positive are eligible if they have received hepatitis B (HBV) antiviral therapy for at least 4 weeks and have undetectable HBV viral load prior to start of trial intervention.

Note: Patients should remain on anti-viral therapy throughout trial intervention and follow local guidelines for HBV anti-viral therapy after completion of trial intervention.

Hepatitis B screening tests are not required unless:

* Known history of HBV infection
* Mandated by local health authority. 12. Patients with a history of hepatitis C (HCV) infection are eligible if HCV viral load is undetectable at screening.

Note: Patients must have completed curative antiviral therapy at least 4 weeks prior to start of trial intervention.

Hepatitis C screening tests are not required unless:

* Known history of HCV infection
* Mandated by local health authority.

Melanoma-specific exclusion criteria:

* Current or prior history of uveal, mucosal, or acral melanoma
* Oligometastatic stage IV melanoma
* History of in-transit metastases within the last 6 months
* Prior therapy targeting BRAF and/or MEK

SCCHN-specific exclusion criteria:

• Nasopharyngeal cancer, unknown primary, nasal cavity or paranasal sinus carcinoma

Exclusion criteria applicable across cohorts:

In addition, patients meeting any of the following criteria must be excluded:

1. Currently participating in or has participated in a trial of an investigational agent or has used an investigational device within 4 weeks of the first dose of trial treatment Note: Patients who have entered the follow-up phase of an investigational trial may participate as long as it has been 4 weeks after the last dose of the previous investigational agent.
2. Any prior treatment for the tumor under study
3. Prior therapy for another tumor with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., CTLA-4, OX40, CD137), and discontinued from that treatment due to a grade 3 or higher immune-related adverse event (irAE)
4. Prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to first dose of trial treatment

   * Note: Patients must have recovered from all adverse events (AEs) due to previous therapies (i.e., grade ≤1 at baseline). Patients with grade ≤2 neuropathy are eligible for the trial. Patients with endocrine-related AEs grade ≤2 requiring treatment or hormone replacement are also eligible.
   * Note: If the patient has had major surgery, the patient must have recovered adequately from the procedure and/or complications from the surgery prior to starting trial treatment.
5. Live or live-attenuated vaccine within 30 days prior to the first dose of trial treatment. Note: Administration of inactivated vaccines, mRNA-based vaccines [e.g., COVID-19] and vector-based vaccines are allowed.
6. Diagnosis of immunodeficiency or receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment. Patients who are currently receiving steroids at a dose equivalent to <5 mg/day of prednisone do not need to discontinue steroids prior to enrollment. Patients who require topical, ophthalmologic and inhalational steroids will not be excluded from the trial. Patients with hypothyroidism stable on hormone replacement or Sjögren's syndrome will not be excluded from the trial.
7. Additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy.
8. History of an allogeneic tissue/solid organ transplant.
9. Active autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Patients with type I diabetes mellitus; hypothyroidism only requiring hormone replacement; skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment; or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
10. History of radiation pneumonitis
11. History of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease
12. Active infection requiring systemic therapy
13. HIV-infected patients with a history of Kaposi sarcoma and/or Multicentric Castleman Disease
14. Has known active hepatitis B virus (HBV; defined as hepatitis B surface antigen [HBsAg] reactive and/or detectable HBV DNA) or known active hepatitis C virus (HCV) (defined as anti HCV Ab positive and detectable HCV ribonucleic acid [RNA] [qualitative]) infection.

    Note: Testing for hepatitis B and hepatitis C is not required unless
    1. Known history of HBV or HCV infection
    2. Mandated by local health authority. Patients with a history of hepatitis will be screened using serology to confirm status.
15. History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the patient's participation for the full duration of the trial, or is not in the best interest of the patient to participate, in the opinion of the treating investigator
16. Psychiatric or substance abuse disorders that would interfere with the patient's ability to cooperate with the trial requirements
17. Severe hypersensitivity (grade ≥3) to pembrolizumab and/or any of its excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-12-21 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Major pathologic response | Observed in the resected tumor tissue after neoadjuvant treatment at surgery
  Major pathologic response, defined as pathologic complete response (pCR) (0% residual viable tumor) or near pCR (≤10% residual viable tumor)

SECONDARY OUTCOMES:
Pathologic complete response | Observed in the resected tumor tissue after neoadjuvant treatment at surgery
  Pathologic complete response (pCR) (0% residual viable tumor)
Pathologic tumor response | Pathologic tumor response of the surgical specimens will be assessed at the time of surgery.
  Pathologic tumor response (≤ 49% residual viable tumor) at surgery
Objective response rate | Determined after 9 weeks of treatment
  Objective response rate (ORR), determined by RECIST 1.1
Disease-free survival | at 2 years after surgery
  Disease-free survival (DFS) from the date of surgery
Event-free survival | Determined after 9 weeks of treatment
  Event-free-survival (EFS)
Event-free survival | at 2 years after surgery
  Event-free-survival (EFS)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Burtness, MD, Prof, Principal Investigator — Yale New Haven Hospital - Yale Cancer Center
Locations (15):
- United States (3):
  - Yale, New Haven, Connecticut
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Massey Cancer Center, Richmond, Virginia
- Australia (2):
  - Melanoma Institute Australia The Uiniversity of Sydney, and Royal North Shore Hospital, Sydney, New South Wales
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
- Denmark (2):
  - Aarhus University Hospital, Aarhus
  - Copenhagen University Hospital Herlev, Copenhagen
- France (3):
  - CHRU Lille, Lille
  - Hôpital Ambroise-Paré, Paris
  - Institut Gustave Roussy, Paris
- Germany (2):
  - Universitätsklinikum Essen & Research Alliance Ruhr, Essen
  - Universität Heidelberg, Medizinische Fakultät, Heidelberg
- Spain (3):
  - Hospital Universitario Quirón Dexeus, Barcelona
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Clínico Universitario de Valencia -INCLIVA, Valencia